CLINICAL TRIAL: NCT03481478
Title: Third Hospital of Hebei Medical University
Brief Title: Detecting Occult Proximal Humeral Neck Fractures Through CT and MRI Tests of Patients With Greater Tuberosity Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HZY2018
Record Dates: First submitted 2018-02-22; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Humeral Greater Tuberosity; Humeral Fractures/ Proximal; Fractures/ Occult
Keywords: occult; proximal humeral neck fractures; greater tuberosity; shoulder dislocation
MeSH Terms: conditions — Shoulder Fractures; Fractures, Closed; Shoulder Dislocation | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with greater tuberosity fractures: If humeral surgical neck fractures can be detected through CT or MRI in such groups.
  Interventions: Diagnostic Test: CT and MRI
- Dislocation patients with greater tuberosity fractures: If humeral surgical neck fractures can be detected through CT or MRI in such groups.
  Interventions: Diagnostic Test: CT and MRI

INTERVENTIONS:
Diagnostic Test: CT and MRI — For such patients, using CT and/or MRI to find if existing humeral surgical neck fractures.

SUMMARY:
Patients with greater tuberosity fractures is becoming increasingly common, as is the number of cases of humeral surgical neck fractures. This study investigated the relationship between size of greater tuberosity fragment and occurrence of humeral surgical neck fractures by using CT or MRI tests.

DETAILED DESCRIPTION:
Some humeral surgical neck fractures can be detected through X-ray of shoulder in patients with greater tuberosity fractures. However, some fractures can not be find through conventional X-ray in such patients unless broader CT or MRI tests are required to confirm diagnoses of humeral surgical neck fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with greater tuberosity fractures and shoulder dislocation/ or not who were acute injured were included

Exclusion Criteria:

* Patients with ipsilateral previous proximal humeral fractures and obviously proximal humeral fractures were excluded。

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient demographics, comorbidities, injury mechanisms and other variables were recorded and calculated for each case.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-24 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Humeral surgical neck fractures can be detected through CT/MRI. | 31/12/2018
  Some greater tuberosity fractures with/or not shoulder dislocation can combined with humeral surgical neck fractures,which can be detected through CT/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Guo Junfei, MD, Study Director — Hebei Medical University Third Hospital
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided